CLINICAL TRIAL: NCT07208526
Title: A Multicenter Randomized Controlled Study on Surgical Decision-Making Guided by the TDTP-RECIST Evaluation System for Locally Advanced Intrahepatic Cholangiocarcinoma Following GOLP Conversion Therapy
Brief Title: A Randomized Trial of Surgical Decision-Making Guided by TDTP-RECIST
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Shanghai Geriatric Medical Center (Other); Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other); Shanghai 10th People's Hospital (Other); Oriental Hepatobiliary Surgery Hospital Affiliated to Naval Military Medical University (Unknown)
Responsible Party: Principal Investigator, Jia Fan, Professor, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZSAB-TDTP-transGOLP
Record Dates: First submitted 2025-09-28; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Intrahepatic Cholangiocarcinoma (Icc); Conversion Therapy; TDTP-RECIST; GOLP Regimen
MeSH Terms: conditions — Cholangiocarcinoma; Cirrhosis, Familial, with Pulmonary Hypertension | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Medication Group (Placebo Comparator): Upon randomization, patients will continue to receive the GOLP regimen for up to 8 cycles, followed by maintenance therapy with lenvatinib plus toripalimab for one year, until disease progression, withdrawal from the study, or the occurrence of intolerable toxicity.
  Interventions: Drug: GOLP regimen
- Surgery Group (Experimental): Surgical resection is to be performed within 2-4 weeks after randomization, followed by adjuvant therapy with capecitabine at a dose of 1250 mg/m² twice daily, administered orally for eight cycles (each cycle consists of 14 days of medication followed by a 7-day rest period, constituting a 3-week treatment cycle).
  Interventions: Procedure: Surgery
- TDTP Group (Experimental): Following randomization, patients will be evaluated using the TDTP-RECIST system. Those who meet the predetermined cutoff value (63%) will proceed to surgical resection. Patients not meeting the cutoff value will continue the GOLP regimen for up to 8 cycles, during which those who subsequently meet the cutoff value will undergo surgery. Postoperative adjuvant therapy will consist of capecitabine (1250 mg/m², BID, orally) for eight cycles (each cycle: 14 days on, 7 days off, constituting a 3-week cycle). Patients who do not meet the cutoff value after 8 cycles of GOLP therapy will receive maintenance therapy with lenvatinib plus toripalimab for up to one year or until intolerable toxicity occurs.
  Interventions: Diagnostic Test: TDTP-RECIST

INTERVENTIONS:
Drug: GOLP regimen — PD1 antibody (Toripalimab) combined with GEMOX chemotherapy and Lenvatinib neoadjuvant treatment
  Arms: Medication Group
Procedure: Surgery — R0 resection
  Arms: Surgery Group
Diagnostic Test: TDTP-RECIST — Treatment selection between continued GOLP therapy and surgical R0 resection based on TDTP-RECIST criteria.
  Arms: TDTP Group

SUMMARY:
This project aims to conduct a prospective, multicenter, randomized controlled clinical trial. The study plans to enroll 270 patients with locally advanced iCCA who have successfully undergone GOLP conversion therapy. Participants will be randomized at a 1:2:2 ratio into three arms: Control Arm (continued medication), Direct Surgery Arm, and TDTP-RECIST Assessment Arm. The primary endpoint is Overall Survival (OS).

DETAILED DESCRIPTION:
Intrahepatic cholangiocarcinoma (iCCA) is a highly aggressive malignancy with a poor prognosis, and a majority of patients are ineligible for curative surgery upon initial diagnosis. Although the GOLP conversion therapy regimen, pioneered by our research team, has demonstrated promising results in preliminary studies-achieving an 80% objective response rate and a 63% R0 resection rate-its clinical value requires validation through high-level evidence-based medicine. Concurrently, the conventional RECIST 1.1 criteria are inadequate for accurately assessing treatment response in iCCA, leading to challenges in surgical decision-making. To address this, we have developed the innovative TDTP-RECIST evaluation system, which preliminary data suggest can more precisely predict surgical opportunities and survival benefits.

This multicenter randomized controlled trial aims to primarily validate the clinical value of the GOLP regimen as conversion therapy for locally advanced intrahepatic cholangiocarcinoma (iCCA), thereby providing high-level evidence-based medical support for its establishment as a standard treatment protocol. Furthermore, the study seeks to verify the efficacy and superiority of the TDTP-RECIST evaluation system in guiding surgical decision-making following conversion therapy for iCCA. The ultimate goals are to establish an individualized treatment pathway based on TDTP-RECIST assessments, optimize the timing of surgery, reduce unnecessary surgical interventions and healthcare resource waste, and consequently offer a reliable decision-making framework for the conversion therapy of locally advanced iCCA. This will provide a precise and powerful tool to facilitate the transition from "unresectable" to "curable" disease.

ELIGIBILITY:
Inclusion Criteria:

-

Subjects eligible to participate in this study must meet all of the following criteria:

1. Male or female aged 18-75 years;
2. Patients must provide signed informed consent prior to enrollment, demonstrating the ability to understand and willingness to sign the written informed consent form;
3. Pathologically confirmed diagnosis of intrahepatic cholangiocarcinoma;
4. Locally advanced disease, failure to achieve R0 resection, and absence of distant metastasis;
5. At least one measurable lesion;
6. Eastern Cooperative Oncology Group (ECOG) performance status score of 0;
7. Child-Pugh class A liver function;

Exclusion Criteria:

-

Subjects who meet any of the following exclusion criteria are not permitted to enroll in this study:

1. Pathologically diagnosed hepatocellular carcinoma, combined hepatocellular-cholangiocarcinoma, or other non-cholangiocarcinoma malignant components;
2. Patients with postoperative recurrence, or those who have previously received PD-1/PD-L1 antibodies, CTLA-4 antibodies, lenvatinib, or chemotherapy;
3. History or current diagnosis of other malignancies;
4. Active tuberculosis infection;
5. Active, known, or suspected autoimmune disease;
6. History of interstitial lung disease, or non-infectious pneumonitis requiring steroid treatment;
7. Significant clinically significant bleeding symptoms within 3 months prior to enrollment, or clear bleeding tendency;
8. Suspected allergy to the investigational drug(s).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 24 months
  the time period from the randomization of the patient to the death event due to any reason

SECONDARY OUTCOMES:
Event-free survival | 24 months
  From randomization to the occurrence of the following events: disease progression prevents radical surgery; local or distant recurrence; second primary tumor; death due to various causes.
Objective response rate | 6 months
  The proportion of patients whose tumor volume has decreased to a predetermined value
Pathological remission rate | 6 months
  the ratio of the estimated active tumor size divided by the tumor bed size
Recurrence-free survival | 24 months
  the time from surgery to disease recurrence or all-cause death
R0 Resection Rate | 12 months
  Curative Surgery Resection Rate
Adverse events | 12 months
  the severity of adverse events will be evaluated according to the NCI CTCAE 5.0 standard

OTHER OUTCOMES:
Exploratory markers | 24 months
  the relationship between treatment response and clinical factors: carcinoembryonic antigen (CEA), carbohydrate antigen 199 (CA199), carbohydrate antigen 125 (CA125), tumor mutation burden (TMB), PD-L1 expression, microsatellite instability (MSI), dynamic changes of PET-CT Standard uptake value, dynamic changes of contrast Ultrasound and MRI

CONTACTS AND LOCATIONS:
Overall Officials: Jia Fan, MD&PhD, Study Chair — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan hospital, Shanghai, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shi G, Huang X, Li X, Liang F, Gao Q, Zhang D, Lu J, Ji Y, Hu Z, Chen Y, Qiu S, Yi Y, Zhu X, Sun H, Shi Y, Peng M, Wang X, Huang C, Ding Z, He Y, Shen Y, Xu Y, Xiao Y, Hu J, Zhou J, Fan J. Conversion therapy of tislelizumab plus lenvatinib and GEMOX in unresectable locally advanced biliary tract cancer (ZSAB-TransGOLP): a multicentre, prospective, phase 2 study. Lancet Oncol. 2025 Oct;26(10):1334-1345. doi: 10.1016/S1470-2045(25)00376-6. Epub 2025 Aug 29. PMID 40889502
- [Background] Shi GM, Huang XY, Wu D, Sun HC, Liang F, Ji Y, Chen Y, Yang GH, Lu JC, Meng XL, Wang XY, Sun L, Ge NL, Huang XW, Qiu SJ, Yang XR, Gao Q, He YF, Xu Y, Sun J, Ren ZG, Fan J, Zhou J. Toripalimab combined with lenvatinib and GEMOX is a promising regimen as first-line treatment for advanced intrahepatic cholangiocarcinoma: a single-center, single-arm, phase 2 study. Signal Transduct Target Ther. 2023 Mar 17;8(1):106. doi: 10.1038/s41392-023-01317-7. PMID 36928584
- [Background] Oh DY, He AR, Bouattour M, Okusaka T, Qin S, Chen LT, Kitano M, Lee CK, Kim JW, Chen MH, Suksombooncharoen T, Ikeda M, Lee MA, Chen JS, Potemski P, Burris HA 3rd, Ostwal V, Tanasanvimon S, Morizane C, Zaucha RE, McNamara MG, Avallone A, Cundom JE, Breder V, Tan B, Shimizu S, Tougeron D, Evesque L, Petrova M, Zhen DB, Gillmore R, Gupta VG, Dayyani F, Park JO, Buchschacher GL Jr, Rey F, Kim H, Wang J, Morgan C, Rokutanda N, Zotkiewicz M, Vogel A, Valle JW. Durvalumab or placebo plus gemcitabine and cisplatin in participants with advanced biliary tract cancer (TOPAZ-1): updated overall survival from a randomised phase 3 study. Lancet Gastroenterol Hepatol. 2024 Aug;9(8):694-704. doi: 10.1016/S2468-1253(24)00095-5. Epub 2024 May 29. PMID 38823398
- [Background] Kelley RK, Ueno M, Yoo C, Finn RS, Furuse J, Ren Z, Yau T, Klumpen HJ, Chan SL, Ozaka M, Verslype C, Bouattour M, Park JO, Barajas O, Pelzer U, Valle JW, Yu L, Malhotra U, Siegel AB, Edeline J, Vogel A; KEYNOTE-966 Investigators. Pembrolizumab in combination with gemcitabine and cisplatin compared with gemcitabine and cisplatin alone for patients with advanced biliary tract cancer (KEYNOTE-966): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2023 Jun 3;401(10391):1853-1865. doi: 10.1016/S0140-6736(23)00727-4. Epub 2023 Apr 16. PMID 37075781
- [Background] Colangelo M, Di Martino M, Polidoro MA, Forti L, Tober N, Gennari A, Pagano N, Donadon M. Management of intrahepatic cholangiocarcinoma: a review for clinicians. Gastroenterol Rep (Oxf). 2025 Jan 26;13:goaf005. doi: 10.1093/gastro/goaf005. eCollection 2025. PMID 39867595
- [Background] Moris D, Palta M, Kim C, Allen PJ, Morse MA, Lidsky ME. Advances in the treatment of intrahepatic cholangiocarcinoma: An overview of the current and future therapeutic landscape for clinicians. CA Cancer J Clin. 2023 Mar;73(2):198-222. doi: 10.3322/caac.21759. Epub 2022 Oct 19. PMID 36260350